CLINICAL TRIAL: NCT06073795
Title: Ultrasound Guided Versus Fluoroscopy Guided Lumber Sympathetic Block in Chronic Lower Limb Ischemia
Brief Title: Ultrasongraphy Versus Fluoroscopy in Lumber Sympathetic Block in Chronic Lower Limb Ischemia
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Sally Ahmed kamel, assistant lecturer, Assiut University
Other Study IDs: sympathetic block in ischemia
Record Dates: First submitted 2023-10-03; First posted 2023-10-10 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: L L Ischemia
MeSH Terms: interventions — Autonomic Nerve Block

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- FL group: Patients will receive FL-guided LSGB with 10 mL of 0.25% bupivacaine.
  Interventions: Procedure: sympathetic block
- US group: Patients will receive US-assisted LSGB with 10 mL of 0.25% bupivacaine.
  Interventions: Procedure: sympathetic block

INTERVENTIONS:
Procedure: sympathetic block — LSGBs will be performed at the lower third of the L2 or the upper third of the L3 vertebra without any premedication. The targeted lumbar vertebra will be identified with an anteroposterior (AP) fluoroscopic imaging in the FL group or with an US longitudinal tracing approach from the caudad to cephalad direction in the US group. The skin entry point will be infiltrated with 1% lidocaine. Then, a curved 21 G, 15-cm Chiba needle will be advanced toward the target using the posterolateral approach in both groups. Each patient will undergo LSGBs according to the allocated group.

SUMMARY:
The aim of this study is to compare total procedure time and success rate between FL-guided and US-assisted LSGBs in Lower Limb Ischemic patients.

DETAILED DESCRIPTION:
Morbidity and death in acute lower limb arterial occlusion are well described. The patients often are in a debilitated state, with multiple concurrent medical comorbidities. An association with hypercoagulable phenomena (e.g., active malignancy) may explain the frequency of some of these conditions. Other conditions, however, may be directly responsible for the occlusive event itself (e.g., the association of myocardial disease and peripheral embolization) (1, 2).

The sympathetic nervous system controls many of the involuntary functions of the human body and plays a role in chronic pain conditions such as complex regional pain syndrome (CRPS) (3).

About 20% of patients who suffered lower limb ischemic pain are not suitable for surgical intervention for various reasons. In these patients, a lumbar sympathetic ganglion block (LSGB) can be used to reduce pain, improve the walking status and activities of daily living, and may delay or avoid amputation. LSGB technique has become increasingly popular in recent decades, and several diseases are treated with LSGB, including neuropathic pain (NP), vascular pain, and erythematous extremity pain (4).

An LSGB refers to injecting drugs (local anesthetic drugs: lidocaine, ropivacaine, etc.) into the lumbar sympathetic ganglia of the corresponding segment to destroy the nerve conduction function, thereby achieving the method of treating certain diseases. The use of LSGB can destroy the innervation of sympathetic nerves on the blood vessels of the lower extremities, and the innervated blood vessels continue to expand to improve local blood circulation and nutrient supply, thereby reducing pain (5).

This block is typically performed in the prone position at the L3 level under fluoroscopic guidance. Fluoroscopy (FL)-guided LSGB has been a popular technique, as it provided great accuracy in confirming the location of needle tip or intravascular (IV) injection. However, this technique exposes patients to radiation and its success rate ranges from 67% with FL guidance to 83% with computed tomography (CT) guidance (6).

Ultrasound (US)-guided or assisted techniques have been introduced to the field of pain medicine in the mid- 2000s. US guidance has been shown to be associated with many advantages, including minimal radiation exposure, as well as the ability to visualize soft tissue structures and observe needle insertion and spread pattern of injectate in real time (7).

As US guidance has undergone technical advancements, its applicability expanded from peripheral blocks to deep neuraxial blocks. A recent technical description of US guidance LSGB in a patient with CRPS type I showed that the anterior fascia of the psoas muscle and the anterolateral part of vertebral body are key landmarks during the procedure (8).

US-guided LSGB in conjunction with FL, may be expected to provide real-time visualization of the needle tip location with respect to the anterior fascia of the psoas major muscle in paravertebral space with an advantage of low radiation exposure.

Recently, numerous US-assisted procedures in pain medicine have been attempted, showing an advantage of low radiation exposure (8).However, only few publications relatively few sample size manipulate the comparison between FL-guided and US-assisted LSGBs in Lower Limb Ischemic patients.

ELIGIBILITY:
Inclusion Criteria:

* • Lower Limb Ischemic patients need LSGB procedures

Exclusion Criteria:

* • A body mass index (BMI) of >30 kg/m2.

  * A history of post-lumbar laminectomy with internal fixation or any severe anatomic variation, such as scoliosis and tumor.
  * History of lumbar sympathetic chemical or thermal neurolysis.
  * Pregnancy.
  * Infection at the puncture site.
  * Coagulopathy.
  * Allergy to local anesthetics.

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Lower Limb Ischemic patients need LSGB procedures
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
the total procedure time | two years
  the time from the first radiographic image for the identification of the lumbar vertebral level to the completion of the bupivacaine injection (FL group), or the time from the US probe placement on the patient's skin to the completion of the bupivacaine injection (US group).

SECONDARY OUTCOMES:
success rate | two years
  measured by vasodilatation which is measured by temperature difference between the limbs
  , imaging time, onset time for temperature rise, bone touching, frequency of needle adjustment, spread pattern of contrast medium, and procedure-related complications.

REFERENCES:
- [Background] Lassandro G, Tamburrini S, Liguori C, Picchi SG, Pezzullo F, Ferrandino G, Spinetti F, Vigliotti G, Marano I, Scaglione M. Lower Limb Ischemia as Acute Onset of Primary Aortic Occlusion: CTA Imaging and Management. Int J Environ Res Public Health. 2023 Feb 22;20(5):3868. doi: 10.3390/ijerph20053868. PMID 36900878
- [Background] Phuphanich ME, Convery QW, Nanda U, Pangarkar S. Sympathetic Blocks for Sympathetic Pain. Phys Med Rehabil Clin N Am. 2022 May;33(2):455-474. doi: 10.1016/j.pmr.2022.02.002. PMID 35526979
- [Background] Awal S, Madabushi R, Agarwal A, Singla V. CRPS: Early Lumbar Sympathetic Block is Better Compared to Other Interventions. Pain Physician. 2016 Feb;19(2):E363. No abstract available. PMID 26815268
- [Background] Samen CDK, Sutton OM, Rice AE, Zaidi MA, Siddarthan IJ, Crimmel SD, Cohen SP. Correlation Between Temperature Rise After Sympathetic Block and Pain Relief in Patients with Complex Regional Pain Syndrome. Pain Med. 2022 Sep 30;23(10):1679-1689. doi: 10.1093/pm/pnac035. PMID 35234922
- [Background] Kanao-Kanda M, Kanda H, Iida T, Kikuchi S, Azuma N. Clinical Application of Laser Speckle Flowgraphy to Assess Changes in Blood Flow to the Foot After a Lumbar Sympathetic Ganglion Block: A Case Report. J Pain Res. 2021 May 26;14:1451-1456. doi: 10.2147/JPR.S305543. eCollection 2021. PMID 34079360
- [Background] Cohen SP, Khunsriraksakul C, Yoo Y, Parker E, Samen-Akinsiku CDK, Patel N, Cohen SJ, Yuan X, Cheng J, Moon JY. Sympathetic Blocks as a Predictor for Response to Ketamine Infusion in Patients with Complex Regional Pain Syndrome: A Multicenter Study. Pain Med. 2023 Mar 1;24(3):316-324. doi: 10.1093/pm/pnac153. PMID 36269190
- [Background] Hurdle MF. Ultrasound-Guided Spinal Procedures for Pain: A Review. Phys Med Rehabil Clin N Am. 2016 Aug;27(3):673-86. doi: 10.1016/j.pmr.2016.04.011. PMID 27468672
- [Background] Ryu JH, Lee CS, Kim YC, Lee SC, Shankar H, Moon JY. Ultrasound-Assisted Versus Fluoroscopic-Guided Lumbar Sympathetic Ganglion Block: A Prospective and Randomized Study. Anesth Analg. 2018 Apr;126(4):1362-1368. doi: 10.1213/ANE.0000000000002640. PMID 29189275